CLINICAL TRIAL: NCT03450811
Title: Does the Inguinal Hernia Repair Affect Uroflowmetric Values? A Prospective Controlled Clinical Trial.
Brief Title: Effect of Inguinal Hernia Repair on Uroflowmetric Parameteres
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Training and Research Hospital (Other)
Collaborators: Ministry of Health, Turkey (Other Government)
Responsible Party: Principal Investigator, Muhammet Fatih Kilinc, Principal investigator, Medical doctor, Ankara Training and Research Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 317
Record Dates: First submitted 2018-02-19; First posted 2018-03-01 (Actual); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Inguinal Hernia; Urinary Retention; Lower Urinary Tract Symptoms
Keywords: complication; uroflowmetry
MeSH Terms: conditions — Hernia, Inguinal; Urinary Retention; Lower Urinary Tract Symptoms

STUDY DESIGN:
Intervention Model Description: The patients who underwent elective open or laparoscopic inguinal hernia repair were treated by a single general surgeon.
Who Masked: Participant
Masking Description: The control group consisted of volunteer participitants who were admitted to the outpatient clinics with various reasons or healthy persons
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Active Comparator): The patients underwent elective open or laparoscopic inguinal hernia repair at a general surgery clinic.
  Interventions: Procedure: Inguinal hernia repair
- Control group (No Intervention): patients who were admitted to the outpatient clinics with various diseases or healthy persons

INTERVENTIONS:
Procedure: Inguinal hernia repair — Lichtenstein procedure or laparoscopic method (Total extraperitoneal) inguinal hernia repair
  Arms: Study group

SUMMARY:
Post operative acute urinary retension or voiding dysfunction are complications after inguinal hernia repair and they cause a great deal of discomfort and stress to patients. Furthermore, they can also increase hospital costs by increasing hospital stay, and by growing the need for outpatient appointments after an elective surgical procedure. Some studies recommend prophylactic alpha blockers to minimizing these adverse effects.

Investigators aimed to determine the changes of uroflowmetric values for male patients following elective inguinal hernia repair.

DETAILED DESCRIPTION:
Inguinal hernia repair is a common procedure performed in general surgery, with an annual rate of 28 per 100,000 of the population in the USA. The incidence of post operative inability voiding in males following open or laparoscopic inguinal hernia repair varies from 3 to 25%. Evaluating risk factors to reduce the occurence of this complications after one of the most commonly performed surgery by general surgeons could help reduce that high rate of that complication. Although some authors recommend prophylactic alpha blockers, there is no consensus on whether these can decrease rate of urinary retention or voiding dysfunction in male patients.

In current study, investigators aimed to determinate the uroflowmetric parametric changes of patients after elective inguinal hernia repair.

ELIGIBILITY:
Inclusion Criteria:

* any type of inguinal hernia

Exclusion Criteria:

* active urinary tract infection,
* previous BPH, neurological disease or significant systemic disease,
* medications that could interfere voiding function
* history of prostate, bladder or urethral surgery or traumatic urethral catheterisation.

Ages: 20 Years to 90 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male patients
Enrollment: 120 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-02-20 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with undergoes inguinal hernia repair -related voiding dysfunction as assessed by uroflowmetry | 3 days
  Maximum and average flow rate (ml/sn) were determinated on post-operative day 1

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Training and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Mohammadi-Fallah M, Hamedanchi S, Tayyebi-Azar A. Preventive effect of tamsulosin on postoperative urinary retention. Korean J Urol. 2012 Jun;53(6):419-23. doi: 10.4111/kju.2012.53.6.419. Epub 2012 Jun 19. PMID 22741052
- [Result] Clancy C, Coffey JC, O'Riordain MG, Burke JP. A meta-analysis of the efficacy of prophylactic alpha-blockade for the prevention of urinary retention following primary unilateral inguinal hernia repair. Am J Surg. 2018 Aug;216(2):337-341. doi: 10.1016/j.amjsurg.2017.02.017. Epub 2017 Mar 14. PMID 28341140